CLINICAL TRIAL: NCT07379827
Title: Effectiveness and Adverse-effect Switch Evaluation
Brief Title: Effectiveness and Adverse-effect Switch Evaluation of Xanomeline and Trospium Chloride (KarXT)
Status: Not yet recruiting | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CN012-0134
Record Dates: First submitted 2026-01-23; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Schizophrenia
Keywords: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — xanomeline; trospium chloride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Participants diagnosed with schizophrenia receiving xanomeline and trospium chloride (KarXT)
  Interventions: Drug: Xanomeline and trospium chloride (KarXT)

INTERVENTIONS:
Drug: Xanomeline and trospium chloride (KarXT) — According to the product label

SUMMARY:
The purpose of this study is to describe real-world treatment patterns, effectiveness and adverse events of adults diagnosed with schizophrenia that have initiated xanomeline and trospium chloride (KarXT) treatment in the United States

ELIGIBILITY:
Inclusion Criteria:

* Participants (or caregiver/legal guardian) must have signed and dated an Institutional Review Board (IRB)/Independent Ethics Committee (IEC)-approved written ICF or signed an electronic ICF in accordance with regulatory, local, and institutional guidelines.
* Adults ≥ 18 years of age at Baseline who are willing and able, in the judgement of the treating clinician, to participate in routine clinical care and follow up.
* Schizophrenia, confirmed by the treating clinician's judgement or physician decision to treat the patient with receiving xanomeline and trospium chloride (KarXT) for schizophrenia made prior to and independently of participation in this study. Current Antipsychotic Treatment: Participant must fall into one of the categories below:

  * Be within <16 weeks of initiating treatment with KarXT with intent to discontinue prior antipsychotic treatment(s) OR
  * On a stable regimen (dose and frequency consistent with the drug label and/or at a stable dose based on the judgement of the Investigator for at least 30 days prior to screening) of treatment with 1 or more antipsychotics with plan to discontinue and switch to treatment with KarXT from a prior antipsychotic treatments(s). NOTE: The decision to switch for reasons of safety, tolerability, and/or efficacy will be made independently by the treating clinician and/or the patient and is not dictated by the study. Participants can be enrolled during tapering/discontinuing process from prior antipsychotic treatment(s). Individuals who are not currently receiving treatment for schizophrenia are not eligible for the study. Any antipsychotic treatments must be recorded as concomitant medications.
* Concomitant psychiatric medications (eg, antidepressants, mood stabilizers, anxiolytics) are permitted and are recommended to remain at a stable dose during the study period.

Exclusion Criteria:

* Prior use of KarXT that has been discontinued for any reason prior to Baseline.
* Participation in an interventional study within the last 30 days or plans to participate in an interventional study at the time of eligibility or baseline through the study period.
* Known hypersensitivity to xanomeline or trospium chloride, or history or high risk of urinary retention, gastric retention, moderate (Child-Pugh Class B) or severe (Child-Pugh Class C) hepatic impairment, or narrow-angle glaucoma.
* In the opinion of the treating clinician, unstable psychiatric or medical conditions that would prevent the participant from safely switching to KarXT. Hospitalized individuals who have been switched to KarXT or are switching treatment to KarXT are permitted to be enrolled at discharge if they are < 16 weeks from initiation of KarXT.
* Participants who are pregnant, planning to become pregnant, or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include adults diagnosed with schizophrenia who have switched or plan to switch from prior antipsychotic treatment to xanomeline and trospium chloride (KarXT)
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Treatment titration and switch regimens as described by the prescribing clinician | Baseline and up to 20 weeks

SECONDARY OUTCOMES:
Adverse events (AEs) | Baseline and up to 20 weeks
Change in participant weight | Baseline and up to 20 weeks
Clinical Global Impressions - Improvement (CGI-I) score | Baseline and up to 20 weeks
Number of schizophrenia-related relapses (defined as schizophrenia-related emergency department visits and/or hospitalizations and symptoms | Baseline and up to 20 weeks
Continuation of treatment with xanomeline and trospium chloride (KarXT) at End of Study | Baseline and up to 20 weeks
Number of participants who discontinue treatment, time to discontinuation, and reasons for discontinuation | Baseline and up to 20 weeks
Number of participants using antiemetic treatment by type, duration, and resolution of event for xanomeline and trospium chloride (KarXT) related gastro-intestinal (GI) symptoms | Baseline and up to 20 weeks
Date of first xanomeline and trospium chloride (KarXT) treatment | Baseline
Participant age | Baseline
Participant sex | Baseline
Participant race | Baseline
Participant ethnicity | Baseline
Participant height | Baseline
Participant's family history of schizophrenia | Baseline
Duration since diagnosis of schizophrenia | Baseline
Previous treatment(s) received for schizophrenia | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Bristol Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- PPD Virtual - PPD - US, Wilmington, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts